CLINICAL TRIAL: NCT00004031
Title: SWOG-9704 A Randomized Phase III Trial Comparing Early High Dose Chemoradiotherapy and an Autologous Stem Cell Transplant to Conventional Dose CHOP Chemotherapy Plus Rituximab for CD20+ B Cell Lymphomas (With Possible Late Autologous Stem Cell Transplant) for Patients With Diffuse Aggressive Non-Hodgkin's Lymphoma in the High-Intermediate and High Risk International Classification Prognostic Groups
Brief Title: SWOG-9704 Chemoradiotherapy and Peripheral Stem Cell Transplantation Compared With Combination Chemotherapy in Treating Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network); Eastern Cooperative Oncology Group (Network); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065658; S9704 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Lymphoma
Keywords: stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult Burkitt lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult Burkitt lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma | interventions — Rituximab; VAP-cyclo protocol; Carmustine; Cyclophosphamide; Doxorubicin; Etoposide; Prednisone; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHOP/CHOP-R x 3 (Active Comparator): Cyclophosphamide 750 mg/m2 IV Day 1 Doxorubicin 50 mg/m2 IV Day 1 Prednisone 100 mg/day PO Days 1-5 Vincristine 1.4 mg/m2 IV Day 1 Rituximab 375 mg/m2 IV Day 1 This regimen is repeated every 21 days for 8 cycles
  Interventions: Biological: rituximab; Drug: CHOP regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate; Procedure: bone marrow ablation with stem cell support
- CHOP/CHOP-R x 1 + Autologous Stem Cell Transplant (Experimental): Cyclophosphamide 750 mg/m2 IV Day 1 Doxorubicin 50 mg/m2 IV Day 1 Prednisone 100 mg/day PO Days 1-5 Vincristine 1.4 mg/m2 IV Day 1 Rituximab 375 mg/m2 IV Day 1 This regimen is repeated every 21 days for 6 cycles followed by autologous stem cell transplant.
  Interventions: Biological: rituximab; Drug: CHOP regimen; Drug: carmustine; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: prednisone; Drug: vincristine sulfate; Procedure: bone marrow ablation with stem cell support; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: rituximab — 375 mg/m2 IV every 21 days
Drug: CHOP regimen
Drug: carmustine
  Arms: CHOP/CHOP-R x 1 + Autologous Stem Cell Transplant
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
  Arms: CHOP/CHOP-R x 1 + Autologous Stem Cell Transplant
Drug: prednisone
Drug: vincristine sulfate
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation
  Arms: CHOP/CHOP-R x 1 + Autologous Stem Cell Transplant
Radiation: radiation therapy
  Arms: CHOP/CHOP-R x 1 + Autologous Stem Cell Transplant

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy and radiation and kill more cancer cells. It is not yet known whether chemoradiotherapy plus peripheral stem cell transplantation is more effective than combination chemotherapy alone in treating non-Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying chemoradiotherapy and peripheral stem cell transplantation to see how well they work compared to combination chemotherapy in treating patients with stage II, stage III, or stage IV non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival and progression-free survival of patients with intermediate- or high-grade non-Hodgkin's lymphoma treated with high-dose chemoradiotherapy and autologous peripheral blood stem cell transplantation (APBSCT) vs conventional dose cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) (or CHOP plus rituximab for CD20+ disease) with possible late APBSCT.
* Compare the toxic effects of these regimens in this patient population.

OUTLINE: This is a randomized study. Patients are stratified according to disease risk (intermediate-high vs high).

Patients receive CHOP chemotherapy comprising cyclophosphamide IV over 15 minutes, doxorubicin IV, and vincristine IV on day 1 and oral prednisone on days 1-5. Patients with CD20-positive disease also receive rituximab IV on day 1 (or day 0 during course 1 only). Treatment repeats every 3 weeks for 5 courses in the absence of disease progression or unacceptable toxicity.

Within 35 days of completing the fifth course, patients with partial or complete response are randomized to one of two treatment arms.

* Arm I: Patients receive CHOP (or CHOP plus rituximab [CHOP-R]) as above. Treatment repeats every 3 weeks for 3 additional courses. After completion of chemotherapy, patients are encouraged to undergo harvest of peripheral blood stem cells (PBSC) for possible use at time of relapse. After completion of 8 courses, patients receive no additional therapy until disease progression or biopsy-proven disease.
* Arm II: Patients receive one additional course of CHOP/CHOP-R followed by filgrastim (G-CSF), sargramostim (GM-CSF), or other colony-stimulating factors used singly or in combination according to center preference. PBSC are harvested and selected for CD34+ cells. Patients under age 61 receive one of two preparative regimens: a total body irradiation (TBI)-based regimen comprising irradiation administered twice daily on days -8 to -5, etoposide IV over 4 hours on day -4, and cyclophosphamide IV over 1 hour on day -2 OR carmustine IV over 2 hours on days -6 to -4 and etoposide and cyclophosphamide as in the TBI-based regimen. Patients age 61 to 65 receive the augmented regimen comprising carmustine, etoposide, and cyclophosphamide as above. Patients receive involved field radiotherapy prior to the preparative regimen only if there is biopsy-proven residual bulk disease and at the discretion of the center. PBSC are reinfused 36-48 hours after completion of cyclophosphamide. If both bone marrow and PBSC are harvested, bone marrow is reinfused on day 0 and then PBSC are reinfused either the same day or the following day.

Patients are followed every 6 months for 2 years and then annually thereafter.

PROJECTED ACCRUAL: Approximately 360 patients (at least 135 per treatment arm) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven intermediate- or high-grade non-Hodgkin's lymphoma
* Ann Arbor classification of "bulky" stage II, III, or IV
* Must be classified as high-intermediate or high-risk according to International Age Adjusted Index
* Bidimensionally measurable disease
* No lymphoblastic, transformed, or mantle cell lymphomas
* No CNS involvement by lymphoma
* CD20 status confirmed by immunocytochemistry or flow cytometry
* Must have either bilateral or unilateral bone marrow aspiration and biopsy ≥ 42 days before first course of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) therapy (or CHOP plus rituximab [CHOP-R] for CD20+ disease) OR within 42 days prior to registration if CHOP/CHOP-R therapy has not begun
* Must have bilateral bone marrow aspiration and biopsy within 28 days of randomization

  * Bone marrow involvement with lymphoma is allowed, provided there is an improvement of at least 50% if used as an evaluable site of disease
* No prior lymphoma, Hodgkin's lymphoma, myelodysplastic syndromes, or leukemia NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 15 to 65

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* No nonlymphoma-related hepatic dysfunction

Renal:

* Creatinine no greater than 2 times ULN
* Creatinine clearance at least 60 mL/min
* No nonlymphoma-related renal dysfunction
* No history of grade 3 hemorrhagic cystitis due to cyclophosphamide

Cardiovascular:

* No coronary artery disease, cardiomyopathy, congestive heart failure, or dysrhythmia requiring therapy
* MUGA scan or 2-D echocardiogram required if patient's history is questionable
* Ejection fraction normal

Pulmonary:

* DLCO or FEV_1 at least 60% of predicted

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No allergy to etoposide
* No active bacterial, fungal, or viral infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior monoclonal antibody therapy for lymphoma except if included in a single course of CHOP/CHOP-R

Chemotherapy:

* No prior chemotherapy for lymphoma except for a single course of CHOP/CHOP-R* NOTE: *Prednisone or other corticosteroids not considered prior chemotherapy

Endocrine therapy:

* See Chemotherapy
* Prior corticosteroids allowed

Radiotherapy:

* No prior radiotherapy for lymphoma
* No prior thoracic radiotherapy or radiotherapy greater than 2,000 cGy to any other site

Surgery:

* Not specified

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 1997-07; Primary Completion 2008-06-01 (Actual); Study Completion 2013-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. Stiff, MD, Study Chair — Loyola University; Thomas C. Shea, MD, Study Chair — UNC Lineberger Comprehensive Cancer Center; David P. Schenkein, MD, Study Chair — Tufts Medical Center Cancer Center; Stephen Couban, MD, Study Chair — Cancer Care Nova Scotia
Locations (15):
- Oregon Health & Science University, Portland, Oregon, United States
- Canada (14):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Moncton Hospital, Moncton, New Brunswick
  - Doctor H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Odette Cancer Centre at Sunnybrook, Toronto, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - Hopital Du Sacre-Coeur de Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Hopital du Saint-Sacrement - Quebec, Québec, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Stiff PJ, Unger JM, Cook J, et al.: Randomized phase III U.S./Canadian intergroup trial (SWOG S9704) comparing CHOP ± R for eight cycles to CHOP ± R for six cycles followed by autotransplant for patients with high-intermediate (H-Int) or high IPI grade diffuse aggressive non-Hodgkin lymphoma (NHL). [Abstract] J Clin Oncol 29 (Suppl 15): A-8001, 2011.
- [Derived] Cook JR, Goldman B, Tubbs RR, Rimsza L, Leblanc M, Stiff P, Fisher R. Clinical significance of MYC expression and/or "high-grade" morphology in non-Burkitt, diffuse aggressive B-cell lymphomas: a SWOG S9704 correlative study. Am J Surg Pathol. 2014 Apr;38(4):494-501. doi: 10.1097/PAS.0000000000000147. PMID 24625415
- [Derived] Stiff PJ, Unger JM, Cook JR, Constine LS, Couban S, Stewart DA, Shea TC, Porcu P, Winter JN, Kahl BS, Miller TP, Tubbs RR, Marcellus D, Friedberg JW, Barton KP, Mills GM, LeBlanc M, Rimsza LM, Forman SJ, Fisher RI. Autologous transplantation as consolidation for aggressive non-Hodgkin's lymphoma. N Engl J Med. 2013 Oct 31;369(18):1681-90. doi: 10.1056/NEJMoa1301077. PMID 24171516

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 397 participants were registered, of whom 27 were ineligible. Of the 370 eligible participants, 117 were excluded from randomization and so only 253 underwent randomization.
Groups:
- CHOP/CHOP-R x 3: Cyclophosphamide 750 mg/m2 IV Day 1 Doxorubicin 50 mg/m2 IV Day 1 Prednisone 100 mg/day PO Days 1-5 Vincristine 1.4 mg/m2 IV Day 1 Rituximab 375 mg/m2 IV Day 1 This regimen is repeated every 21 days for 8 cycles
  rituximab: 375 mg/m2 IV every 21 days
  CHOP regimen
  cyclophosphamide
  doxorubicin hydrochloride
  prednisone
  vincristine sulfate
  bone marrow ablation with stem cell support
- CHOP/CHOP-R x 1 + Autologous Stem Cell Transplant: Cyclophosphamide 750 mg/m2 IV Day 1 Doxorubicin 50 mg/m2 IV Day 1 Prednisone 100 mg/day PO Days 1-5 Vincristine 1.4 mg/m2 IV Day 1 Rituximab 375 mg/m2 IV Day 1 This regimen is repeated every 21 days for 6 cycles followed by autologous stem cell transplant.
  rituximab: 375 mg/m2 IV every 21 days
  CHOP regimen
  carmustine
  cyclophosphamide
  doxorubicin hydrochloride
  etoposide
  prednisone
  vincristine sulfate
  bone marrow ablation with stem cell support
  peripheral blood stem cell transplantation
  radiation therapy
Period: Overall Study
Arm/Group | CHOP/CHOP-R x 3 | CHOP/CHOP-R x 1 + Autologous Stem Cell Transplant
Started | 128 | 125
Assessed for Adverse Events | 123 | 113
Completed | 103 | 104
Not Completed | 25 | 21
Not completed — Adverse Event | 5 | 0
Not completed — Refusal unrelated to adverse events | 2 | 11
Not completed — Progression/relapse | 9 | 4
Not completed — Death | 3 | 1
Not completed — Other- not protocol specified | 3 | 3
Not completed — Reason under review | 3 | 2

BASELINE CHARACTERISTICS:
Population: Eligible participants that were randomized to study arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | CHOP/CHOP-R x 3 | CHOP/CHOP-R x 1 + Autologous Stem Cell Transplant | Total
Number analyzed (Participants) | 128 | 125 | 253
Age, Continuous [Median (Full Range); unit: years] | 51.3 [19.8 to 65.8] | 49.6 [18.5 to 66.2] | 50.6 [18.5 to 66.2]
Age, Customized [Number; unit: percentage of participants]
  % >=60 years | 18 | 20 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 49 | 105
  Male | 72 | 76 | 148
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 113 | 106 | 219
  Unknown or Not Reported | 13 | 15 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 6 | 7 | 13
  White | 119 | 109 | 228
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4
WHO B Cell Histology [Count of Participants; unit: Participants]
  WHO B Cell Histology | 114 | 110 | 224
  Diffuse Large B-Cell,Not Otherwise Specified | 78 | 86 | 164
WHO T Cell Histology [Count of Participants; unit: Participants]
  WHO T Cell Histology | 14 | 15 | 29
  Peripheral T, Not otherwise Specified | 4 | 6 | 10
Immunophenotyping [Count of Participants; unit: Participants]
  B cell CHOP-R | 76 | 75 | 151
  B cell CHOP | 40 | 35 | 75
Stage [Count of Participants; unit: Participants] — Staging based on the Ann Arbor staging criteria and on extent of disease at the time of diagnosis. Bulky disease determination made after surgical resection.
  Stage II: involvement of 2 or more lymph nodes on same side of diaphragm or localized involvement of an extralymphatic organ or site
  Stage III: lymph nodes on both sides of diaphragm which may be accompanied by localized involvement of an extralymphatic organ or site
  Stage IV: diffuse or disseminated involvement of one or more extralymphatic organs with/without associated lymph node or isolated extralymphatic organ involvement
  Participants
    Bulky II | 9 | 4 | 13
    III | 3 | 44 | 47
    IV | 78 | 78 | 156
Performance status >= 2 [Count of Participants; unit: Participants] — Participants were graded according to the SWOG grading scale
  2: Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more that 50% of waking hours
  3: Capable of only limited self-care; confined to bed or chair more than 50% of waking hours.
  4: Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  5: Dead
  Participants | 44 | 48 | 92
Elevated LDH [Count of Participants; unit: Participants] — Serum LDH greater than institutional upper limit of normal
  Participants | 104 | 106 | 210
B Symptoms [Count of Participants; unit: Participants] — Staging based on the Ann Arbor staging criteria
  B symptoms- fever, sweats, weight loss > 10% of body weight
  Participants | 81 | 75 | 156
International Prognostic Index: High [Count of Participants; unit: Participants] — Number of risks factors (stage III or IV disease, serum LDH greater than normal, performance status of 2-4) participants have.
  High-Intermediate risk: 2 risk factors High risk: 3 risk factors
  Participants | 44 | 44 | 88
Extra nodal Sites >=2 [Count of Participants; unit: Participants] | 29 | 31 | 60
Bone marrow involvement- Yes [Count of Participants; unit: Participants] — Presence of lymphoma in the bone marrow based off of bone marrow biopsy done within 42 days prior to the first cycle of therapy
  Participants | 31 | 19 | 50

OUTCOME MEASURES:

1. Primary Outcome: 2-year Overall Survival Rates
Description: Percentage of participants surviving 2 years post registration
Time Frame: up to 2 years post registration
Population: Eligible participants that were randomized to study arms.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CHOP/CHOP-R x 3 | CHOP/CHOP-R x 1 + Autologous Stem Cell Transplant
Number analyzed (Participants) | 128 | 125
percentage of participants | 71.1 [63.2 to 78.9] | 73.7 [66.0 to 81.4]

2. Primary Outcome: 2 Year Progression-free Survival
Description: Percentage of participants without disease progression up to 2 years post-registration.
Time Frame: From registration until death
Population: Eligible participants that were randomized to study arms.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CHOP/CHOP-R x 3 | CHOP/CHOP-R x 1 + Autologous Stem Cell Transplant
Number analyzed (Participants) | 128 | 125
percentage of participants | 55.4 [46.9 to 64.1] | 69.1 [61.0 to 77.1]

3. Secondary Outcome: Number of Patients With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE Version 2.0. Only adverse events that are possibly, probably or definitely related to study drug are reported.
  Higher grades indicate higher severity of adverse events.
Time Frame: Duration of treatment and follow up until death or 3 years post registration
Population: Patients who received at least one dose of protocol treatment.
Measure: Number; unit: Participants
Groups:
- CHOP/CHOP-R x 3: Cyclophosphamide 750 mg/m2 IV Day 1 Doxorubicin 50 mg/m2 IV Day 1 Prednisone 100 mg/day PO Days 1-5 Vincristine 1.4 mg/m2 IV Day 1 Rituximab 375 mg/m2 IV Day 1 This regimen is repeated every 21 days for 8 cyclesXXrituximab: 375 mg/m2 IV every 21 daysXXCHOP regimenXXcyclophosphamideXXdoxorubicin hydrochlorideXXprednisoneXXvincristine sulfateXXbone marrow ablation with stem cell support
- CHOP/CHOP-R x 1 + Autologous Stem Cell Transplant: Cyclophosphamide 750 mg/m2 IV Day 1 Doxorubicin 50 mg/m2 IV Day 1 Prednisone 100 mg/day PO Days 1-5 Vincristine 1.4 mg/m2 IV Day 1 Rituximab 375 mg/m2 IV Day 1 This regimen is repeated every 21 days for 6 cycles followed by autologous stem cell transplant.XXrituximab: 375 mg/m2 IV every 21 daysXXCHOP regimenXXcarmustineXXcyclophosphamideXXdoxorubicin hydrochlorideXXetoposideXXprednisoneXXvincristine sulfateXXbone marrow ablation with stem cell supportXXperipheral blood stem cell transplantationXXradiation therapy
Arm/Group | CHOP/CHOP-R x 3 | CHOP/CHOP-R x 1 + Autologous Stem Cell Transplant
Number analyzed (Participants) | 123 | 113
Participants
  Abdominal pain/cramping | 8 | 9
  Alkaline phosphatase increase | 9 | 15
  Allergic reaction | 0 | 8
  Allergic rhinitis | 4 | 5
  Alopecia | 43 | 36
  Anemia | 57 | 89
  Anorexia | 8 | 32
  Anxiety/agitation | 2 | 12
  Apnea | 0 | 1
  Arthralgia | 5 | 15
  Arthritis | 0 | 1
  Ataxia (incoordination) | 2 | 6
  Bicarbonate decrease | 0 | 1
  Bilirubin increase | 3 | 6
  Blurred vision | 0 | 4
  Bone pain | 6 | 4
  Bruising | 0 | 2
  CO diffusion capacity decrease | 0 | 2
  Cardiac ischemia/infarction | 0 | 1
  Cardiovascular-other | 0 | 4
  Catheter related infection | 1 | 11
  Chest pain,not cardio or pleur | 4 | 9
  Colitis | 0 | 2
  Confusion | 1 | 5
  Conjunctivitis | 0 | 1
  Constipation/bowel obstruction | 14 | 24
  Cough | 15 | 32
  Creatinine increase | 2 | 7
  Cushingoid appearance | 0 | 1
  Dehydration | 3 | 7
  Delusions | 0 | 1
  Depression | 3 | 12
  Diarrhea without colostomy | 13 | 49
  Dizziness/light headedness | 9 | 8
  Dizziness/vertigo, NOS | 1 | 1
  Double vision | 1 | 1
  Dry skin | 1 | 4
  Dyspepsia/heartburn | 6 | 10
  Dyspnea | 17 | 26
  Dysuria | 1 | 2
  Ear-other | 1 | 0
  Earache | 0 | 1
  Edema | 9 | 32
  Endocrine-other | 0 | 1
  Epistaxis | 0 | 4
  Erectile impotence | 0 | 2
  Eryth/rash/eruption/desq, NOS | 1 | 2
  Erythema multiforme/blistering | 0 | 1
  Esophagitis/dysphagia | 3 | 9
  Eye-other | 0 | 1
  FEV1 decrease | 0 | 3
  Fatigue/malaise/lethargy | 47 | 67
  Febrile neutropenia | 10 | 44
  Fever without neutropenia | 5 | 17
  Fever, NOS | 5 | 5
  Flu-like symptoms-other | 0 | 2
  Flushing | 1 | 18
  Focal dermatitis | 0 | 2
  GGT increase | 0 | 1
  GI Mucositis, NOS | 1 | 10
  GI-other | 0 | 2
  GU-other | 0 | 1
  GVHD | 0 | 3
  Gastritis | 0 | 2
  Gynecomastia | 1 | 0
  Hallucinations | 0 | 2
  Hand-foot skin reaction | 1 | 3
  Headache | 6 | 26
  Hematuria | 0 | 4
  Hemorrhage-other | 1 | 5
  Hiccoughs | 0 | 6
  Hot flashes | 3 | 3
  Hyperglycemia | 4 | 21
  Hyperkalemia | 0 | 1
  Hypermagnesemia | 0 | 1
  Hypernatremia | 0 | 2
  Hypertension | 0 | 5
  Hyperuricemia | 2 | 2
  Hypoalbuminemia | 1 | 10
  Hypocalcemia | 1 | 13
  Hypoglycemia | 0 | 1
  Hypokalemia | 2 | 10
  Hypomagnesemia | 0 | 6
  Hyponatremia | 2 | 9
  Hypophosphatemia | 0 | 9
  Hypotension | 1 | 15
  Hypoxia | 0 | 6
  Infection w/o 3-4 neutropenia | 4 | 13
  Infection with 3-4 neutropenia | 6 | 17
  Infection, unk ANC | 0 | 2
  Inner ear-hearing loss | 0 | 2
  Insomnia | 9 | 15
  Invol. movement/restlessness | 0 | 2
  Joint,muscle,bone-other | 4 | 0
  Keratitis | 0 | 1
  LVEF decrease/CHF | 2 | 3
  Leukopenia | 68 | 81
  Liver-other | 1 | 0
  Local injection site reaction | 1 | 0
  Lung-other | 1 | 2
  Lymphedema | 1 | 0
  Lymphopenia | 59 | 80
  Melena/ GI bleeding | 1 | 2
  Memory loss | 2 | 0
  Menses changes | 1 | 3
  Metabolic-other | 0 | 1
  Mouth dryness | 1 | 9
  Muscle weakness (not neuro) | 4 | 10
  Myalgia | 15 | 19
  Myalgia/arthralgia, NOS | 2 | 4
  Nail changes | 3 | 2
  Nausea | 31 | 66
  Neuro-other | 1 | 2
  Neuropathic pain | 1 | 1
  Neutropenia/granulocytopenia | 60 | 89
  PRBC transfusion | 3 | 32
  Pain-other | 15 | 17
  Palpitations | 0 | 2
  Partial thromboplast time inc | 1 | 5
  Pericar. effusion/pericarditis | 0 | 1
  Personality/behavioral change | 1 | 0
  Petechiae/purpura | 0 | 2
  Phlebitis | 3 | 0
  Pigmentation changes/yellowing | 3 | 3
  Platelet transfusion | 2 | 37
  Pleural effusions | 1 | 3
  Pneumonitis/infiltrates | 2 | 10
  Proctitis | 0 | 2
  Proteinuria | 0 | 1
  Prothrombin time increase | 1 | 3
  Pruritus | 3 | 7
  Pulmonary edema | 0 | 1
  Pulmonary fibrosis | 0 | 1
  RT-GI mucositis, NOS | 0 | 2
  RT-esophagitis | 0 | 1
  RT-focal dermatitis, NOS | 0 | 1
  RT-pain | 0 | 1
  RT-pharyngeal dysphagia | 0 | 2
  Rash/desquamation | 7 | 35
  Rectal bleeding/hematochezia | 0 | 2
  Rectal/anal fistula | 0 | 1
  Rectal/perirectal pain | 0 | 3
  Renal failure | 0 | 1
  Reportable adverse event, NOS | 1 | 0
  Respiratory infect w/ neutrop | 0 | 3
  Respiratory infect w/o neutrop | 4 | 3
  Respiratory infection, unk ANC | 0 | 1
  Rigors/chills | 2 | 15
  SGOT (AST) increase | 9 | 15
  SGPT (ALT) increase | 2 | 9
  SIADH | 0 | 1
  Salivary gland changes | 0 | 3
  Second primary | 1 | 0
  Sense of smell | 0 | 2
  Sensory neuropathy | 46 | 40
  Sinus bradycardia | 2 | 4
  Sinus tachycardia | 2 | 12
  Skin-other | 3 | 6
  Somnolence/consciousness loss | 0 | 2
  Stomatitis/pharyngitis | 12 | 57
  Supraventricular arrhythmia | 0 | 3
  Surgery-wound infection | 0 | 1
  Sweating | 9 | 11
  Syncope | 1 | 0
  Syndrome-other | 0 | 3
  Taste disturbance | 7 | 16
  Thrombocytopenia | 15 | 61
  Thrombosis/embolism | 3 | 3
  Transplant-diarrhea | 0 | 3
  Transplant-granulocytopenia | 0 | 5
  Transplant-leukopenia | 0 | 11
  Transplant-pRBC transfusion | 1 | 1
  Transplant-plt transfusion | 1 | 3
  Transplant-rash/desquamation | 0 | 3
  Transplant-stomatitis/pharyng | 0 | 1
  Transplant-thrombocytopenia | 0 | 13
  Tremor | 0 | 1
  Urinary electrolyte wasting | 0 | 1
  Urinary frequency/urgency | 1 | 3
  Urinary retention | 0 | 1
  Urinary tr infect w/ neutrop | 0 | 1
  Urinary tr infect w/o neutrop | 2 | 2
  VOD associated weight gain | 0 | 1
  Vaginal bleeding | 0 | 2
  Vaginal dryness | 0 | 1
  Vaginitis | 0 | 3
  Vision,NOS | 0 | 1
  Voice change/stridor/larynx | 0 | 1
  Vomiting | 15 | 40
  Weakness (motor neuropathy) | 13 | 4
  Weight gain | 7 | 8
  Weight loss | 2 | 11

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 3 years post registration
Description: Of 253 eligible participants, 17 did not receive protocol therapy so were not assessed for AEs. Therefore only 236 participants were assessed for AEs.
Arm/Group | CHOP/CHOP-R x 3 | CHOP/CHOP-R x 1 + Autologous Stem Cell Transplant
All-Cause Mortality (participants affected / at risk) | 51/128 | 39/125
Serious Adverse Events (participants affected / at risk) | 4/123 | 4/113
Other Adverse Events (participants affected / at risk) | 108/123 | 106/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CHOP/CHOP-R x 3 (N=123) | CHOP/CHOP-R x 1 + Autologous Stem Cell Transplant (N=113)
LVEF decrease/CHF (Cardiac disorders) | 1 | 0
Stomatitis/pharyngitis (Gastrointestinal disorders) | 0 | 1
Reportable adverse event, NOS (General disorders) | 1 | 0
Syndrome-other (General disorders) | 0 | 1
Infection with 3-4 neutropenia (Infections and infestations) | 1 | 0 — Infection with grade 3-4 neutropenia [present or life-threatening sepsis (e.g., septic shock)]
Second primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis/infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CHOP/CHOP-R x 3 (N=123) | CHOP/CHOP-R x 1 + Autologous Stem Cell Transplant (N=113)
Anemia (Blood and lymphatic system disorders) | 57 | 89
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 44
PRBC transfusion (Blood and lymphatic system disorders) | 3 | 32
Platelet transfusion (Blood and lymphatic system disorders) | 2 | 37
Sinus tachycardia (Cardiac disorders) | 2 | 12
Abdominal pain/cramping (Gastrointestinal disorders) | 8 | 9
Constipation/bowel obstruction (Gastrointestinal disorders) | 14 | 24
Diarrhea without colostomy (Gastrointestinal disorders) | 13 | 49
Dyspepsia/heartburn (Gastrointestinal disorders) | 6 | 10
Esophagitis/dysphagia (Gastrointestinal disorders) | 3 | 9
GI Mucositis, NOS (Gastrointestinal disorders) | 1 | 10
Mouth dryness (Gastrointestinal disorders) | 1 | 9
Nausea (Gastrointestinal disorders) | 31 | 66
Stomatitis/pharyngitis (Gastrointestinal disorders) | 12 | 56
Vomiting (Gastrointestinal disorders) | 15 | 40
Edema (General disorders) | 9 | 32
Fatigue/malaise/lethargy (General disorders) | 47 | 67
Fever without neutropenia (General disorders) | 5 | 17
Pain-other (General disorders) | 15 | 17
Rigors/chills (General disorders) | 2 | 15
Sweating (General disorders) | 9 | 11
Allergic reaction (Immune system disorders) | 0 | 8
Infection w/o 3-4 neutropenia (Infections and infestations) | 4 | 13
Infection with 3-4 neutropenia (Infections and infestations) | 5 | 17
Catheter related infection (Injury, poisoning and procedural complications) | 1 | 11
Alkaline phosphatase increase (Investigations) | 9 | 15
Bilirubin increase (Investigations) | 3 | 6
Creatinine increase (Investigations) | 2 | 7
Leukopenia (Investigations) | 68 | 81
Lymphopenia (Investigations) | 59 | 80
Neutropenia/granulocytopenia (Investigations) | 60 | 89
SGOT (AST) increase (Investigations) | 9 | 15
SGPT (ALT) increase (Investigations) | 2 | 9
Thrombocytopenia (Investigations) | 15 | 61
Transplant-leukopenia (Investigations) | 0 | 11
Transplant-thrombocytopenia (Investigations) | 0 | 13
Weight gain (Investigations) | 7 | 8
Weight loss (Investigations) | 2 | 11
Anorexia (Metabolism and nutrition disorders) | 8 | 32
Dehydration (Metabolism and nutrition disorders) | 3 | 7
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 21
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 10
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 13
Hypokalemia (Metabolism and nutrition disorders) | 2 | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 6
Hyponatremia (Metabolism and nutrition disorders) | 2 | 9
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 15
Chest pain,not cardio or pleur (Musculoskeletal and connective tissue disorders) | 4 | 9
Muscle weakness (not neuro) (Musculoskeletal and connective tissue disorders) | 4 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 19
Ataxia (incoordination) (Nervous system disorders) | 2 | 6
Dizziness/light headedness (Nervous system disorders) | 9 | 8
Headache (Nervous system disorders) | 6 | 26
Sensory neuropathy (Nervous system disorders) | 46 | 40
Taste disturbance (Nervous system disorders) | 7 | 16
Weakness (motor neuropathy) (Nervous system disorders) | 13 | 4
Anxiety/agitation (Psychiatric disorders) | 2 | 12
Depression (Psychiatric disorders) | 3 | 12
Insomnia (Psychiatric disorders) | 9 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 32
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 | 26
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Pneumonitis/infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 43 | 36
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 7
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7 | 35
Skin-other (Skin and subcutaneous tissue disorders) | 3 | 6
Flushing (Vascular disorders) | 1 | 18
Hypotension (Vascular disorders) | 1 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No